CLINICAL TRIAL: NCT03443167
Title: RCParvulari: Knowledge, Attitudes and Practices on Cardiopulmonary Resuscitation (CPR) in the Infant Population.
Brief Title: Cardiopulmonary Resuscitation by Children
Acronym: RCParvulari
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Principal Investigator, David Pedrazas, Principal Investigator, Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 4R17/094
Record Dates: First submitted 2018-01-31; First posted 2018-02-23 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Cardiopulmonary Arrest With Successful Resuscitation
Keywords: Cardiopulmonary Resuscitation; Teaching Material; Primary education

STUDY DESIGN:
Intervention Model Description: multicentric clinical trial based on an ad hoc questionnaire
Who Masked: Outcomes Assessor
Masking Description: Only the phase of data analysis will be masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Training on emergency telephone numbers and mnemonics
  Interventions: Behavioral: Training on emergency telephone numbers and mnemonics
- Control group (Sham Comparator): Sham generic formation on the cardiopulmonary arrest.
  Interventions: Behavioral: Sham generic formation on the cardiopulmonary arrest.

INTERVENTIONS:
Behavioral: Training on emergency telephone numbers and mnemonics — The intervention will consist in carrying out an initial theoretical training on how to act in case of attending an emergency, with graphic support of slides (power-point) during 5 minutes, followed by a practical part with the projection of the video of a song and with a "role play" activity for 15 minutes, to remember the helpline number for emergencies (112) and relate it to the mnemonic mouth-nose-eyes. At the beginning and at the end of the theoretical-practical activity, the evaluation questionnaires will be administered to each one of the students.
  Arms: Intervention group
Behavioral: Sham generic formation on the cardiopulmonary arrest. — The sham intervention for the control group will consist in providing a generic formation on the cardiopulmonary arrest, with graphic support of slides (power-point) during 10 minutes, without specifying the telephone number of assistance for emergencies or the mnemonics mouth-nose-eyes. At the beginning and at the end of the theoretical activity, the evaluation questionnaires will be administered to each one of the students.
  Arms: Control group

SUMMARY:
Children's education students are able to identify a possible emergency and in their case act appropriately.

The authors think that the propsed training will improve the knowledge, change the attitude and improve their practical skills, and also retain the information over time.

DETAILED DESCRIPTION:
Cardiopulmonary Resuscitation (CPR) formation in children and teachers is a current and high impact topic in public health: with an appropriate training anyone can save life (Böttiger, 2015). Primary school students are willing to learn CPR and they are also Carriers of knowledge among their surroundings like family or friends (Martínez, 2015).

The authors propose a clinical trial to evaluate the knowledge, attitudes and skills in primary education students of various schools, before and after a CPR formation.

The schools will be previously randomized in intervention group and control group. Once the intervention has been completed and the results obtained, training equal to the intervention will be offered to the control schools. In the bibliographic search no validated questionnaires in CPR learning among primary education students has been found.

ELIGIBILITY:
Inclusion Criteria:

* Spanish primary education students attending the 5th level.
* Informed consent signed by parents or tutors

Exclusion Criteria:

• Spanish primary school children with learning disabilities.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1327 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Learning the helpline number for emergencies (112). | baseline
  Number of children who know the helpline number for emergencies (112),through ad hoc questionnaire, at baseline before and after intervention or sham formation.

SECONDARY OUTCOMES:
Learnig the relatinoship between helpline number for emergencie to the mnemonic mouth-nose-eyes | baseline
  Number of children who know the relatinoship between helpline number for emergencies to the mnemonic mouth-nose-eyes, through ad hoc questionnaire, at baseline before and after intervention or sham formation.
Improvement or maintenance of the knowledge of the helpline number for emergencies (112) | 6-12 months
  Number of children who mantain or improve the knowledge of the helpline number for emergencies (112), through ad hoc questionnaire, after 6-12 months
Improvement or maintenance of the knowledge of the relatinoship between helpline number for emergencie to the mnemonic mouth-nose-eyes | 6-12 months
  Number of children who who mantain or improve the knowledge of the relatinoship between helpline number for emergencie to the mnemonic mouth-nose-eyes, through ad hoc questionnaire, after 6-12 months

CONTACTS AND LOCATIONS:
Overall Officials: David Pedrazas, PhD, Principal Investigator — Institut Català de la Salut. Jordi Gol i Gurina Foundation
Locations (1):
- Abrera, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bottiger BW, Van Aken H. Kids save lives--Training school children in cardiopulmonary resuscitation worldwide is now endorsed by the World Health Organization (WHO). Resuscitation. 2015 Sep;94:A5-7. doi: 10.1016/j.resuscitation.2015.07.005. Epub 2015 Jul 21. No abstract available. PMID 26209417
- [Background] Martínez Villegas I, Varo Caro MC, Salado Natera MI. Metodología didáctica para la en-señanza de reanimación cardiopulmonar en edad infantil. Med Gen y Fam. 2015;4(2):43-46.
- See also: Martínez I 2015: Children are also carriers of knowledge among their surroundings like family or friends — http://www.elsevier.es/es-revista-medicina-general-familia-edicion-digital--231-sumario-vol-4-num-2-S1889543315X0003X